CLINICAL TRIAL: NCT00993005
Title: Efficacy of CICATRIX (Asian Gotu Kola or Pennywort) in the Treatment of Hypertrophic Scars and Keloids Scars.
Brief Title: CICATRIX in the Treatment of Hypertrophic Scars and Keloids Scars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Alfredo Abreu Daniel, "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0910-CU
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Hypertrophic Scars; Keloids
Keywords: Hypertrophic scars; Keloids; Asian Gotu Kola; Asian Pennywort
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid | interventions — Cosmetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Cicatrix
  Interventions: Other: Cicatrix
- B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Cicatrix — Dosage commensurate with surface to be treated. After washing and drying the affected area, a thin layer of CICATRIX (Topical use) will be applied on the scar rubbing in different directions for 2 minutes, three times a day, for 12 weeks.
  Other Names: Cosmetic
  Arms: A
Other: Placebo — Dosage commensurate with surface to be treated. After washing and drying the affected area, a thin layer of PLACEBO (Topical use) will be applied on the scar rubbing in different directions for 2 minutes, three times a day, for 4 weeks.
  Arms: B

SUMMARY:
The purpose of the study is to assess the efficacy of CICATRIX (Asian Gotu Kola or Pennywort) usage in the treatment of Hypertrophic scars and keloids. The duration of this double-blind placebo controlled phase 3 clinical trial will be 12 weeks. The estimated number of persons to be recruited and randomized for the study is 90.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic wound or keloid with no treatment for more than 1 month.
* Signed informed consent.

Exclusion Criteria:

* Usage of steroids within 30 days.
* Malignant neoplastic conditions.
* Alcoholism.
* Handicap and/or psychiatric condition preventing treatment accomplishment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Length of the hypertrophic scar(s) and keloids measured by a millimetric ruler at week 12 (end of the treatment) | 12 weeks

SECONDARY OUTCOMES:
Occurrence of adverse effects at week 12 (end of the treatment) | 12 weeks
Photographs of lesions at week 12 (end of the treatment) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omara Lemus, MD, Principal Investigator — "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital
Locations (1):
- "Cdte. Manuel Fajardo Rivero" Clinical-Surgical-Docent Hospital, Havana, La Habana, Cuba